CLINICAL TRIAL: NCT03060837
Title: To Investigate the Effect of Reducing Renal Movement by Single Lung Ventilation in Patients Administered Retrograde Infrarenal Surgery (RIRS) for Kidney Stones on Operative and Postoperative Parameters
Brief Title: Investigate the Renal Movement by Single Lung Ventilation in Patients Administered RIRS for Kidney Stones.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Boran, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 17
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Perioperative/Postoperative Complications; Kidney Stone
Keywords: RIRS; Kidney Stone; Single lung ventilation; Simultaneous normal ventilation
MeSH Terms: conditions — Postoperative Complications; Kidney Calculi | interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients given single lung ventilation (Active Comparator): The first group will have single lung ventilation applied to ensure reduction. Preoperative Parameters : Hmg, serum creatinine levels Peroperative Parameters : Scope duration, perforation, hemorrhage, etc. complications) Postoperative parameters (stone-free rates, complications like postoperative hemorrhage and fever, hospital stay, etc) Movement of kidney : Changes in renal stone position during simultaneous normal ventilation and single lung ventilation.
  Interventions: Diagnostic Test: Preoperative Parameters; Other: Peroperative Parameters; Other: Postoperative Parameters; Other: Movement of kidney; Procedure: single lung ventilation
- Patients given standard ventilation (Active Comparator): This group will have standard ventilation. Preoperative Parameters : Hmg, serum creatinine levels Peroperative Parameters : Scope duration, perforation, hemorrhage, etc. complications) Postoperative parameters (stone-free rates, complications like postoperative hemorrhage and fever, hospital stay, etc) Movement of kidney : Changes in renal stone position during simultaneous normal ventilation and single lung ventilation.
  Interventions: Diagnostic Test: Preoperative Parameters; Other: Peroperative Parameters; Other: Postoperative Parameters; Other: Movement of kidney; Procedure: standard ventilation

INTERVENTIONS:
Diagnostic Test: Preoperative Parameters — Preoperative Hmg and serum creatinine levels
Other: Peroperative Parameters — Scope duration, perforation, hemorrhage, etc. complications
Other: Postoperative Parameters — Stone-free rates, complications like postoperative hemorrhage and fever, hospital stay, etc
Other: Movement of kidney — Changes in renal stone position during simultaneous normal ventilation and single lung ventilation.
Procedure: single lung ventilation — Patients in this group will intubated with an endotracheal tube and then a bronchial blocker will be placed with the help of a fiberoptic bronchoscope or will be intubated with a double lumen endobronchial tube. One lung ventilation will be applied
  Arms: Patients given single lung ventilation
Procedure: standard ventilation — Patients in this group will be intubated with standart single lumen endotracheal tubes and standart two lung ventilation will be applied.
  Arms: Patients given standard ventilation

SUMMARY:
In patients undergoing RIRS for kidney stone, we aim to show the effect of single lung ventilation with a double lumen tube on operative (operation scope duration, perforation, hemorrhage, etc. complications) and postoperative parameters (stone-free rates, complications like postoperative hemorrhage and fever, hospital stay, etc.) and to show changes in renal stone position during simultaneous normal ventilation and single lung ventilation.

DETAILED DESCRIPTION:
In recent years open surgical treatment has changed to minimal invasive treatments for kidney stone treatment. Additionally, the treatment choices vary depending on the localization of the stone and its dimensions. In the European Urology Association (EUA) guidelines, it states the RIRS method can be used to treat stones up to 2 cm in the kidney. Due to RIRS the operation and scopy durations and hospital stay have clearly reduced compared to the standard treatment of percutaneous nephrolithotomy. However, the high hydrostatic pressure applied to the renal pelvis during RIRS may cause unwanted results in the postoperative period such as hydronephrosis and loss of renal parenchyma. During the operation, the stone may move during deep inspirium and expirium sequences linked to deep ventilation which may lengthen the operation and scope durations and brings risks such as perforation during laser lithotripsy application. In this study we aimed to apply single lung ventilation during the operation (one of the indications for single lung ventilation is to increase surgical view and ease manipulation) to minimize renal movement on that side and reduce peroperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years
2. ASA (American Society of Anesthesiologists) 1-3
3. Patients with 2-3 cm stones in kidneys

Exclusion Criteria:

1. Patients with staghorn stones in kidneys
2. Patients with urinary system anomalies

Removal Criteria :

1. Difficult airway
2. Patients with carinal, bronchial lesions
3. Patients with bad general situation
4. Patients younger than 18 years
5. Satiated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in renal stone position during ventilation | 1-2 Hours
  During the operation, the stone may move during deep inspirium and expirium sequences linked to deep ventilation which may lengthen the operation. Preoperative and postoperative Scope will be used to evolve the renal movement. The values will be recorded in milimeters by comparing it.

SECONDARY OUTCOMES:
Scope duration | 10-30 Seconds
  Movement of the kidney during the procedure may cause peroperative complications and lengthen operation and scope durations.
Total anesthesia duration | 1-2 Hours
  Movement of the kidney during the procedure may cause peroperative complications and lengthen operation and scope durations.
Hospital stay | 1-3 Days
  During the operation, the stone may move during deep inspirium and expirium sequences linked to deep ventilation which may lengthen the operation and scope durations and brings risks such as perforation during laser lithotripsy application. It may effect hospital stay duration.

OTHER OUTCOMES:
Perop-postop complications | 1-2 Days
  Single lung ventilation during the operation (one of the indications for single lung ventilation is to increase surgical view and ease manipulation) to minimize renal movement on that side and reduce peroperative and postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Faruk Boran, Study Chair — Kahramanmaraş Üniversitesi
Locations (1):
- Kahramanmaraş Sütçü Imam Üniversity, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No